CLINICAL TRIAL: NCT06628167
Title: Community Support Program for Lung Cancer Screening Volume II
Acronym: LCS II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 08524
Record Dates: First submitted 2024-08-26; First posted 2024-10-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Transportation; Appointments and Schedules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- West Philadelphia (Experimental): Eligible patient population lives in West Philadelphia
  Interventions: Behavioral: Transportation; Behavioral: Scheduling
- Southwest Philadelphia (No Intervention): Eligible patient population lives in Southwest Philadelphia

INTERVENTIONS:
Behavioral: Transportation — Participants with ordered low dose CT and participants with scheduled low dose CT are offered free transportation to and from appointment. Participants with ordered low dose CT are also offered assistance in connecting with scheduling staff.
  Arms: West Philadelphia
Behavioral: Scheduling — Participants with ordered low dose CT are offered assistance in connecting with scheduling staff.
  Arms: West Philadelphia

SUMMARY:
This is a West Philadelphia based community project to improve adherence to lung cancer screening. The overall objective of this project is to demonstrate the impact of a community support program (CSP) on improve adherence to LCS follow-up guidelines in an urban environment. The study will target individuals in the Penn Medicine healthcare system residing in Philadelphia with an upcoming or missed follow-up screening or orders placed but who have not yet scheduled their screenings by offering free transportation coordination to and from the appointment. The study team will also offer to connect those with placed but unscheduled low dose CT orders to connect with Penn Medicine's scheduling staff.

ELIGIBILITY:
Inclusion Criteria:

* Upcoming or missed low dose CT for lung cancer screening
* Philadelphia resident

Exclusion Criteria:

* Lives outside Philadelphia city limits

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Measure the impact of the community support program in improving adherence to lung cancer screening follow-up | 6 months
  The study will measure the impact of a CSP on a population level by using aggregated neighborhood level data. The database has records of patients who had baseline LCS with individual level residential address geocoded to determine neighborhood. West Philadelphia planning district is the intervention group because it's within the catchment area of Penn Medicine, has the highest number of LCS patients, and has consistent high rates of smoking and lung cancer mortality. The control group is patients from Southwest Philadelphia planning district which has a similar Yost score: composite index of socioeconomic status.
  The study will compare the rate of appointment attendance between West Philadelphia patients with scheduled/ordered LCS (intervention group), and appointment attendance of Southwest Philadelphia patients with scheduled/ordered LCS. The study will measure if there's a significant difference made by a CSP on a patient's likelihood of LCS attendance.

CONTACTS AND LOCATIONS:
Overall Officials: Farouk Dako, MD, Principal Investigator — farouk.dako@pennmedicine.upenn.edu
Locations (1):
- Univeristy of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT06628167/ICF_000.pdf